CLINICAL TRIAL: NCT06019013
Title: A Phase 1 Study to Evaluate the Safety and Efficacy Investigate the Immunogenicity and Pharmacokinetic Characteristics of QLF3108 Injection in Patients With Advanced Solid Tumors
Brief Title: A Study of QLF3108 in Participants With Advanced Solid Tumor
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QLF3108-101
Record Dates: First submitted 2023-08-23; First posted 2023-08-31 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose-Escalation Stage and PK-Expansion Stage (Experimental): Dose-Escalation Stage：Participants will be assigned sequentially to escalating doses of QLF3108, up to the maximum tolerated dose (MTD).
  PK-Expansion Stage：1-4 recommended expansion dose will be proposed for the PK-expansion stage of the trial.
  Interventions: Drug: QLF3108

INTERVENTIONS:
Drug: QLF3108 — QLF3108 will be administered independent of body weight.

SUMMARY:
This study will evaluate the safety, tolerability, pharmacokinetics, and immunogenicity of QLF3108 and will make a preliminary assessment of the anti-tumor activity of QLF3108 in patients with advanced solid tumor.

DETAILED DESCRIPTION:
This is a single-arm, open-label, Phase 1, dose escalation and Pharmacokinetics (PK) expansion study of QLF3108 in subjects with advanced solid tumor, to determine the dose-limiting toxicity (DLT), the maximum tolerated dose (MTD) and establish a recommended Phase 2 dose (RP2D) of QLF3108. The purpose of this study is to describe the safety and tolerability, assess pharmacokinetics parameters and immunogenicity, and assess the anti-tumor activity of QLF3108 in subjects with advanced solid tumor.

ELIGIBILITY:
Inclusion Criteria:

1. The volunteer has fully given informed consent to the study and voluntarily signed the informed consent form prior to trial.
2. ≥18 years old and body weight ≥40 kg; Female or male.
3. Histologically or cytologically documented advanced solid tumor;
4. Failed to standard therapy or intolerance, or lack standard therapy advanced solid tumors.
5. Eastern Cooperative Oncology Group（ECOG） performance status of 0 or 1.
6. Life expectancy of at least 12 weeks.
7. Adequate hematologic and end organ function.
8. Female subjects who are not pregnant or not breastfeeding. A negative blood pregnancy test for females of childbearing potential within 7 days prior to first dosing.
9. Male and female subjects of childbearing potential must agree to use highly effective method of contraception during the entire course of the study and within 180 days after the end of the study.

Exclusion Criteria:

1. Patients that have previously received cancer therapy within 4 weeks prior to the first dose of the investigational drug.
2. Patient has received other investigational drug or other clinical trial treatment within 4 weeks prior to the first dose of the investigational drug.
3. Active autoimmune disease that has required systemic treatment within 2 years prior to this study.
4. A live vaccine or live attenuated vaccine was administered within 30 days prior to the first dose of the investigational drug.
5. Patients with Adverse Events(AEs) from previous treatment that have not recovered to ≤1(CTCAE 5.0）; or are unstable status.
6. Severe concomitant medical condition for bowel obstruction, or implanted colon stent during screening period.
7. Patients with a history of HIV positive or other immunodeficiency. Or patients with the history of organ transplant or allogeneic bone marrow (excluding corneal transplantation).
8. Patients with a history of psychiatric disorders, or epilepsy or dementia, drug or alcohol abuse, may impact patient completion of the study.
9. Patients may interfere with the interpretation of study results as determined by the investigator, or are unable to participate in the whole study, or deemed unsuitable by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2023-08-16 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
DLTs of QLF3108 | Approximately 24 months
  dose-limiting toxicity
MTD(s) of QLF3108 | Approximately 24 months
  the maximum tolerated dose
RP2D of QLF3108 | Approximately 24 months
  a recommended Phase 2 dose

SECONDARY OUTCOMES:
The number, rates and severity of participants with Treatment-emergent Adverse Events (TEAEs) according to NCI-CTCAE V5.0 | Approximately 24 month
  The number, rates and severity of participants with Treatment-emergent Adverse Events (TEAEs) according to NCI-CTCAE V5.0
The number, rates and severity of participants with Serious Adverse Events (SAEs) according to NCI-CTCAE V5.0 | Approximately 24 month
  The number, rates and severity of participants with Serious Adverse Events (SAEs) according to NCI-CTCAE V5.0
Cmax of QLF3108 | Approximately 24 month
  Pharmacokinetics of QLF3108 by assessment of maximum plasma QLF3108 concentration.
Tmax of QLF3108 | Approximately 24 month
  Pharmacokinetics of QLF3108 by assessment of time to Cmax
Area under the plasma concentration-time curve (AUC) of QLF3108 | Approximately 24 month
  Pharmacokinetics of QLF3108 by assessment of area under the plasma concentration time curve from zero to infinity
Tl/2 of QLF3108 | Approximately 24 month
  Pharmacokinetics of QLF3108 by assessment of the terminal half-life
Overall Response Rate (ORR) | Approximately 24 months
  ORR is defined as the proportion of patients with a complete response (CR) or partial response (PR) as determined by the investigator according to Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1)
Duration of Response (DOR) | Approximately 24 months
  DOR defined as the time from the first occurrence of a documented objective response to disease progression or death from any cause (whichever occurs first), as determined by the investigator according to RECIST v1.1
Progression-free survival (PFS) | Approximately 24 months
  PFS defined as the time from baseline to first observed disease progression or death from any cause
Overall survival time (OS) | Approximately 24 months
  Overall survival (OS) is the time between the subject's first infusion QLF3108 injection and death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Xu Jianming, M.D, Principal Investigator — Chinese People's Liberation Army (PLA) General Hospital
Locations (1):
- Chinese People's Liberation Army (PLA) General Hospital, Beijing, Beijing Municipality, China